CLINICAL TRIAL: NCT06983314
Title: Prescription Patterns of Antidepressants, Analgesics, and Antiepileptics Drugs in Adult Patients With Acquired Brain Injury Hospitalized in Rehabilitation Center Following Acute Care: a Bicentric Retrospective Study
Brief Title: Prescription Patterns of Antidepressants, Analgesics, and Antiepileptics Drugs in Adult With Acquired Brain Injury
Acronym: PRES'SMR
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 4726
Record Dates: First submitted 2025-02-03; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-01

CONDITIONS: Acquired Brain Injury Including Stroke
Keywords: Acquired Brain Injury; Stroke; Traumatic Brain Injury; Rehabilitation; Prescription Patterns; Antidepressants; Antiepileptics; Analgesics; Drug Complications; Adverse Drug Reactions; Drug-Drug Interactions; Pharmacological Management; Post-acute Care
MeSH Terms: conditions — Brain Injuries; Stroke; Brain Injuries, Traumatic; Drug-Related Side Effects and Adverse Reactions | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: Patients with Acquired Brain Injury (ABI) receiving prescribed antidepressants, antiepileptics, and analgesics during hospitalization.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of pharmacological prescriptions in patients with ABI

SUMMARY:
Acquired brain injury (ABI), primarily caused by stroke and traumatic brain injury (TBI), leads to severe disabilities and requires complex pharmacological management during post-acute rehabilitation. The lack of dedicated guidelines and regular treatment re-evaluation increases the risk of adverse drug reactions (ADRs).

Retrospective, bicentric study in two rehabilitation centers in Normandy, France, from November 1, 2020, to October 31, 2023, to describe prescription patterns of antidepressants, antiepileptics, and analgesics, as well as potential drug-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Adults hospitalized in a rehabilitation center for acquired brain injury (ABI) after passing through an acute care department.
* ABI must be the primary diagnosis in the PMSI (French medical information system).
* The pharmacological classes of interest (antidepressants, antiepileptics, analgesics) must have been introduced during acute care or within the first month of hospitalization in the rehabilitation center.

Exclusion Criteria:

* Patients who did not receive new prescriptions for the pharmacological classes of interest during acute care or the first month of hospitalization in the rehabilitation center.
* Patients who were already prescribed these drugs prior to the ABI.
* Patients who were not hospitalized immediately after discharge from acute care (patients must have been transferred directly from acute care to the rehabilitation center, without spending time in another department or at home).
* Patients who were transferred to an emergency department during rehabilitation and did not return to the rehabilitation center.
* Patients who died during hospitalization or were discharged against medical advice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with acquired brain injury (ABI) who were hospitalized in two rehabilitation centers in Normandy, France, between November 1, 2020, and October 31, 2023. Eligible patients were required to have passed through an acute care department before being admitted to the rehabilitation center. Only patients with ABI as the primary diagnosis, according to the PMSI (French medical information system), were included.
  The study focused on patients who received new prescriptions for specific pharmacological classes (antidepressants, antiepileptics, and analgesics) either during acute care or within the first month of rehabilitation hospitalization. Patients were excluded if they had pre-existing prescriptions for these drugs prior to ABI, or if they did not receive new prescriptions for these drugs during the study period.
  The final study population was selected based on these inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Prescription Paterns and rates of antidepressants, antiepileptics and analgesics | From the date of admission to the rehabilitation center to the date of discharge from the rehabilitation center (median duration of stay approximately 100 days).
  Proportion of patients with at least one prescription of antidepressants, antiepileptics, or analgesics retrieved from medical records, described at three time points: (1) pre-existing usual prescriptions prior to acute care hospitalization, (2) prescriptions at discharge from acute care, and (3) prescriptions at discharge from rehabilitation.
  This outcome is purely descriptive. No clinical events are measured. No measurement tools are used. Data are extracted retrospectively from medical records.

SECONDARY OUTCOMES:
Total number of drugs listed per prescription type | From the date of admission to the rehabilitation center to the date of discharge from the rehabilitation center (median duration of stay approximately 100 days).
  To analyze the average number of drugs per prescription, categorized into three types: usual prescription, discharge from acute care, and discharge from rehabilitation.
  Unit of Measure:
  Number of drugs per prescription Retrieval of prescriptions of interest from the medical file, analysis and data collection. No use of measurement tool. Just description of prescriptions.
Most frequently prescribed drug classes per prescription type | From the date of admission to the rehabilitation center to the date of discharge from the rehabilitation center (median duration of stay approximately 100 days).
  To identify the top prescribed pharmacological classes (e.g., using ATC classification) within usual prescriptions, acute discharge prescriptions, and rehabilitation discharge prescriptions.
  Unit of Measure:
  Number of prescriptions per drug class Retrieval of prescriptions of interest from the medical file, analysis and data collection. No use of measurement tool. Just description of prescriptions.
Analysis of specific drugs, their indications, and therapeutic management | From the date of admission to the rehabilitation center to the date of discharge from the rehabilitation center (median duration of stay approximately 100 days)
  To describe the most frequently prescribed drugs in the three target classes, assess whether their indications comply with official labelling, and detail any therapeutic adjustments during the rehabilitation stay (e.g., dosage changes, discontinuation).
  Unit of Measure:
  Number of prescriptions assessed for compliance and change Retrieval of prescriptions of interest from the medical file, analysis and data collection. No use of measurement tool. Just description of prescriptions.
Number of potential drug-drug interactions identified | From the date of admission to the rehabilitation center to the date of discharge from the rehabilitation center (median duration of stay approximately 100 days).
  To identify and count potential pharmacokinetic or pharmacodynamic drug-drug interactions involving antidepressants, antiepileptics, or analgesics, in the context of all prescribed medications.
  Unit of Measure:
  Number of potential drug-drug interactions per patient Retrieval of prescriptions of interest from the medical file, analysis and data collection. No use of measurement tool. Just description of prescriptions.
Rate of suspected Adverse Drug Reactions (ADRs) and therapeutic consequences | From the date of admission to the rehabilitation center to the date of discharge from the rehabilitation center (median duration of stay approximately 100 days).
  To identify suspected Adverse Drug Reactions (ADRs) reported in medical records and describe the related clinical decisions (e.g., discontinuation, switch, dose adjustment).
  Unit of Measure:
  Number of ADRs reported and management decisions documented Retrieval of prescriptions of interest from the medical file, analysis and data collection. No use of measurement tool. Just description of prescriptions.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen (Centre Hospitalier Universitaire de Caen, France), Caen, France

IPD SHARING:
Plan to Share IPD: No